CLINICAL TRIAL: NCT03558477
Title: A Dose Blocked-randomized, Open-label, Parallel Design Clinical Trial to Assess the Pharmacokinetic/Pharmacodynamic Properties and Safety of YYD601 After Oral Administration in Healthy Adult Male Volunteers(Phase 1)
Brief Title: PK/PD Clinical Trial of YYD601 in Healthy Adult Male
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YYPCT_YYD601_P1
Record Dates: First submitted 2017-10-11; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Intervention Model Description: Each arm is assignted 10 persons[the percent of each arm is (treatmnet: comparator=4:1)]
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Set 1(YYD601 1 & Nexium) (Experimental): Set 1: YYD601 1 & Nexium
  Interventions: Drug: YYD601 1; Drug: Nexium
- Set 2(YYD601 2 & Nexium) (Experimental): Set 2: YYD601 2 & Nexium
  Interventions: Drug: YYD601 2; Drug: Nexium
- Set 3(YYD601 3 & Nexium) (Experimental): Set 3:YYD601 3 & Nexium
  Interventions: Drug: YYD601 3; Drug: Nexium

INTERVENTIONS:
Drug: YYD601 1 — YYD601 1
  Arms: Set 1(YYD601 1 & Nexium)
Drug: YYD601 2 — YYD601 2
  Arms: Set 2(YYD601 2 & Nexium)
Drug: YYD601 3 — YYD601 3
  Arms: Set 3(YYD601 3 & Nexium)
Drug: Nexium — Nexium

SUMMARY:
A dose block-randomized, open-label, parallel clinical trial

DETAILED DESCRIPTION:
This study to evaluate comparatively a characteristics and safety of the PK/PD of single/repeated oral administration YYD601 and Nexium tab and the effects of food influence the PK/PD of YYD601 in healthy adult male.

ELIGIBILITY:
Inclusion criteria:

* Healthy adult male above 19 years old when getting a screening test.
* Subjects who have over 50kg weight, included in the IBW± 20% range. [IBW(kg)={height(cm)-100}x0.9
* Subjects who haven't any congenital or chronic disease, and any other disease following the medical examination.
* Subjects who are confirmed as a participant by the serum test, hematologital test, blood chemistry tests, urine tests, and clinical laboratory test, 12-lead EKG etc following the characteristics aboht the IP within the 3 weeks before investogator products are administrated.
* Subjects who voluntarily decide to participated in this trial after comletely understand about this clinical trial.

Exclusion criteria

* Subjects who are judged not suitable to participated in this trial.
* Other specific exlusion criteria is identified in the protocol.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — healthy adult male
Enrollment: 30 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
half-life | Evaluate the before/after treatment period(5 days per phase)
  Blood sampling time: 1d, 5d, 12d, 16d(each 17 times) half-life(after single dose), (after repeated dose)
Tmax | Evaluate the before/after treatment period(5 days per phase)
  Blood sampling time: 1d, 5d, 12d, 16d(each 17 times) Tmax(after singlidose), Tmax.ss(after repeated dose)
Concentration | Evaluate the before/after treatment period(5 days per phase)
  Blood sampling time: 1d, 5d, 12d, 16d(each 17 times) Cmax(after singlidose), Cmax.ss(after repeated dose) Cmin.ss(after single dose),Cmin.ss(after single dose)
AUC | Evaluate the before/after treatment period(5 days per phase)
  Blood sampling time: 1d, 5d, 12d, 16d(each 17 times) AUClast(after singlidose), AUCt(after repeated dose) AUCinf(after single dose), AUCinf(after repeated dose)

SECONDARY OUTCOMES:
Percent of pH>4 duration time | Evaluate the before/after treatment period(5 days per phase)
  pH>4 duration time
% change in serum gastrin level | Evaluate the before/after treatment period(5 days per phase)
  serum gastrin level

OTHER OUTCOMES:
Adverse event monitoring check up the adverse events | Evaluate the before/after treatment period(5 days per phase)
  Adverse events
Adverse event monitoring check up the vital sign(blood-pressure, pulse rate, temparature) | Evaluate the before/after treatment period(5 days per phase)
  vital sign(blood-pressure, pulse rate, temparature)
Adverse event monitoring check up the 12-lead EKG | Evaluate the before/after treatment period(5 days per phase)
  12-lead EKG
Adverse event monitoring check up the clinical laboratory test | Evaluate the before/after treatment period(5 days per phase)
  clinical laboratory test
Adverse event monitoring check up the physical | Evaluate the before/after treatment period(5 days per phase)
  physical
Adverse event monitoring check up the administraton about the combined drugs | Evaluate the before/after treatment period(5 days per phase)
  administraton about the combined drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungpook national university hospital, Daegu, South Korea

REFERENCES:
- [Derived] Lee HW, Kang WY, Jung W, Gwon MR, Cho K, Yoon YR, Seong SJ. Pharmacokinetics and Pharmacodynamics of YYD601, a Dual Delayed-Release Formulation of Esomeprazole, Following Single and Multiple Doses in Healthy Adult Volunteers Under Fasting and Fed Conditions. Drug Des Devel Ther. 2022 Mar 6;16:619-634. doi: 10.2147/DDDT.S338131. eCollection 2022. PMID 35281316